CLINICAL TRIAL: NCT02809612
Title: The EMBLA Project - An Internet-based Intervention as a Supplement to Clinical Management for Vulvodynia Patients
Brief Title: An Internet-based Information Platform for Vulvodynia Patients
Acronym: EMBLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMBLA
Record Dates: First submitted 2016-03-09; First posted 2016-06-22 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Vulvodynia
MeSH Terms: conditions — Vulvodynia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet-based intervention (Experimental): Patients randomized to the internet-based intervention will be given access to the information in the internet-based platform directly after randomization. During the first 6 weeks, information will be offered in a structured way, with a "theme" changing weekly. After this time-point, the patients will have the possibility to navigate through all information. The platform encompasses internet-based training including information on the disorder, psycho-education and information of simple self-implemented intervention strategies cope with vulvodynia and ameliorate dyspareunia. The platform will also include videos where team members will describe their role in treating patients with the disorder, but also short videos from former patients willing to share their individual stories.
  Interventions: Behavioral: Internet-based platform
- Control group (No Intervention): Patients randomized to the control group through the platform will immediately be informed about the fact that there is available information and resources on the internet and that they will be called for a visit to the physiotherapist-midwife at due time, according to the present guidelines of care followed in the respective clinic (Uppsala, Falun, Gävle).

INTERVENTIONS:
Behavioral: Internet-based platform — Internet-based platform with information and training modules based on acceptance and commitment therapy for vulvodynia patients
  Arms: Internet-based intervention

SUMMARY:
Vulvodynia is a very common but vastly under-diagnosed and under-treated gynaecological condition that leads to extreme suffering for both the women involved but also their partners. It has also been shown to be associated with poor quality of life, leading to depression and anxiety states. When left untreated, the condition takes a very long time to resolve, with a substantial associated disability and suffering. Both psycho-education and internet-based interventions have been shown to be highly successful while they can be quite affordable. This makes them highly cost-effective. The present study aims at evaluating the effectiveness of such an intervention among a vulvodynia patient population from the clinics of Uppsala, Falun, Orebro and Gävle. The patients will be recruited by treating physicians and given access to the internet-based platform, where they will fill out questionnaires during four different time-points, after randomization to the control or the intervention group. The intervention group will also have access to multiple activities and information material uploaded in the internet-based platform. Differences in pain, quality of life and mental health parameter outcomes will be assessed at the end of the study. Should this intervention prove effective, it will be implemented in clinical praxis in the four regions.

ELIGIBILITY:
Inclusion Criteria:

* Vulvodynia patients at their initial evaluation visit to a physician providing written informed consent for participation in the study

Exclusion Criteria:

* inability to read and understand Swedish
* severe mental illness
* currently in treatment for vulvodynia

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Unprovoked pain change, post-intervention | Baseline to post-intervention (6 weeks)
  Change in self-reported unprovoked pain assessment, assessed by Visual Analogue Scale (VAS), between baseline and post-intervention (6 weeks)
Unprovoked pain change, end of clinical treatment | Baseline to end of clinical treatment (typically 10-12 months) or 1 year following inclusion
  Change in self-reported unprovoked pain assessment, assessed by Visual Analogue Scale (VAS), between baseline and after completion of clinical treatment or 1 year following inclusion.
Unprovoked pain change, one year post-treatment | 1 year after end of clinical treatment
  Change in self-reported unprovoked pain assessment, assessed by Visual Analogue Scale (VAS), between baseline and 1 year after completion of clinical treatment.
Provoked pain change, post-intervention | post-intervention (6 weeks)
  Change in self-reported provoked pain assessment, assessed by Visual Analogue Scale (VAS), between baseline and post-intervention (6 weeks)
Provoked pain change, end of clinical treatment | after clinical treatment (typically 10-12 months) or 1 year following inclusion
  Change in self-reported provoked pain assessment, assessed by Visual Analogue Scale (VAS), between baseline and after completion of clinical treatment or 1 year following inclusion.
Provoked pain change, one year post-treatment | 1 year after ending of clinical treatment
  Change in self-reported unprovoked pain assessment, assessed by Visual Analogue Scale (VAS), between baseline and 1 year after completion of clinical treatment.

SECONDARY OUTCOMES:
Satisfaction with Life change | Baseline to post-intervention (6 weeks)
  Change in satisfaction with Life, assessed with Satisfaction with Life Scale, between baseline and post-intervention (6 weeks)
Sexuality | Baseline to post-intervention (6 weeks)
  Change in sexuality measures, assessed by Female Sexual Function Index (FSFI)
Number of visits for clinical treatment | One year after the end of clinical treatment
  Number of visits for clinical treatment
Cost-effectiveness, assessed with the EQ-5D scale | Baseline to one year after completion of clinical treatment
  Cost-effectiveness, assessed with the EQ-5D scale, from baseline to one year after completion of clinica treatment
Sexual function parameters | Baseline to end of clinical treatment
  Change in sexual function parameters, assessed by the Female Sexual Dysfunction Scale (SFDS), between baseline and completion of clinical treatment
Number of days off work | Baseline to end of clinical treatment
Satisfaction with Life change, one year post-treatment | Baseline to one year post-treatment
  Change in satisfaction with Life, assessed with Satisfaction with Life Scale, between baseline and one year after completion of clinical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Alkistis Skalkidou, MD, PhD, Principal Investigator — Dept of Women's and Children's Health, Uppsala University
Locations (1):
- Gynecological Department, Akademiska Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haefner HK. Report of the International Society for the Study of Vulvovaginal Disease terminology and classification of vulvodynia. J Low Genit Tract Dis. 2007 Jan;11(1):48-9. doi: 10.1097/01.lgt.0000225898.37090.04. No abstract available. PMID 17194952
- [Background] Arnold LD, Bachmann GA, Rosen R, Rhoads GG. Assessment of vulvodynia symptoms in a sample of US women: a prevalence survey with a nested case control study. Am J Obstet Gynecol. 2007 Feb;196(2):128.e1-6. doi: 10.1016/j.ajog.2006.07.047. PMID 17306651
- [Background] Harlow BL, Stewart EG. A population-based assessment of chronic unexplained vulvar pain: have we underestimated the prevalence of vulvodynia? J Am Med Womens Assoc (1972). 2003 Spring;58(2):82-8. PMID 12744420
- [Background] Haefner HK, Collins ME, Davis GD, Edwards L, Foster DC, Hartmann ED, Kaufman RH, Lynch PJ, Margesson LJ, Moyal-Barracco M, Piper CK, Reed BD, Stewart EG, Wilkinson EJ. The vulvodynia guideline. J Low Genit Tract Dis. 2005 Jan;9(1):40-51. doi: 10.1097/00128360-200501000-00009. PMID 15870521
- [Background] Amstadter AB, Broman-Fulks J, Zinzow H, Ruggiero KJ, Cercone J. Internet-based interventions for traumatic stress-related mental health problems: a review and suggestion for future research. Clin Psychol Rev. 2009 Jul;29(5):410-20. doi: 10.1016/j.cpr.2009.04.001. Epub 2009 Apr 7. PMID 19403215
- [Background] Tursi MF, Baes Cv, Camacho FR, Tofoli SM, Juruena MF. Effectiveness of psychoeducation for depression: a systematic review. Aust N Z J Psychiatry. 2013 Nov;47(11):1019-31. doi: 10.1177/0004867413491154. Epub 2013 Jun 5. PMID 23739312
- [Background] Backman H, Widenbrant M, Bohm-Starke N, Dahlof LG. Combined physical and psychosexual therapy for provoked vestibulodynia-an evaluation of a multidisciplinary treatment model. J Sex Res. 2008 Oct-Dec;45(4):378-85. doi: 10.1080/00224490802398365. PMID 18937129
- [Background] Bohm-Starke N. Medical and physical predictors of localized provoked vulvodynia. Acta Obstet Gynecol Scand. 2010 Dec;89(12):1504-10. doi: 10.3109/00016349.2010.528368. PMID 21080898
- [Background] Heddini U, Bohm-Starke N, Nilsson KW, Johannesson U. Provoked vestibulodynia--medical factors and comorbidity associated with treatment outcome. J Sex Med. 2012 May;9(5):1400-6. doi: 10.1111/j.1743-6109.2012.02665.x. Epub 2012 Feb 29. PMID 22376009
- [Background] Desrochers G, Bergeron S, Khalife S, Dupuis MJ, Jodoin M. Provoked vestibulodynia: psychological predictors of topical and cognitive-behavioral treatment outcome. Behav Res Ther. 2010 Feb;48(2):106-15. doi: 10.1016/j.brat.2009.09.014. Epub 2009 Oct 7. PMID 19879555
- [Background] Wijma B, Wijma K. A Cognitive Behavioral Treatment Model of Vaginismus. Scand J Behav Ther 1997;26:147-156.
- [Background] Palm A, Danielsson I. SFOGs ARG-rapport för tonårsgynekologi. Sexuell och reproduktiv hälsa hos ungdomar 2013:73-76.
- [Background] Chapple CR, Zimmern PE, Brubaker L, Smith ARB, Bo K. Multidisciplinary Management of Female Pelvic Floor Disorders. Philadelphia: Churchill Livingstone Elsevier; 2006.
- [Derived] Hess Engstrom AH, Kullinger M, Jawad I, Hesselman S, Buhrman M, Hogberg U, Skalkidou A. Internet-based treatment for vulvodynia (EMBLA) - Study protocol for a randomised controlled study. Internet Interv. 2021 Apr 20;25:100396. doi: 10.1016/j.invent.2021.100396. eCollection 2021 Sep. PMID 33996511
- Available data/document: Study Protocol — http://www.kbh.uu.se